CLINICAL TRIAL: NCT02194166
Title: An Open-Label, Randomized, Cross-Over, Multicenter, Phase IIIb Study, to Assess Patients' Tolerability of Trastuzumab Administrated Subcutaneously (SC) Either Via a Single Use Injection Device (SID) or Via Vial for Manual Administration (SC Vial) in Patients With HER2-Positive Early Breast Cancer (eBC)
Brief Title: A Study to Investigate the Tolerability of Subcutaneous (SC) Trastuzumab Administration in Participants With Human Epidermal Growth Factor Receptor 2 (HER2) Positive Early Breast Cancer (eBC) Using Either a Single-Use Injection Device or Manual Administration
Acronym: ESCAPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML28839
Record Dates: First submitted 2014-07-08; First posted 2014-07-18 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Docetaxel

ARMS (3):
- Pre-Randomization (Trastuzumab IV) (Experimental): Trastuzumab IV will be given during the first 4 cycles for all participants before randomization for SC administration. A dose of 6 milligrams per kilogram (mg/kg) will be given every 3 weeks. All the participants will require a loading dose on Day 1 of Cycle 1, so they will receive 8 mg/kg followed by 6 mg/kg, 3 weeks later and then 3-weekly. Concurrent administration during the first 4 cycles of trastuzumab IV with paclitaxel/docetaxel will have to be performed in accordance with local hospital practice.
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: Docetaxel
- Group A: Trastuzumab SC (First Vial Formulation, then SID) (Experimental): Participants will receive 7 cycles of SC trastuzumab 600 mg with assisted administration using a conventional syringe and needle (SC vial formulation) followed by 7 cycles of SC trastuzumab 600 mg SID administration after cross-over.
  Interventions: Drug: Trastuzumab
- Group B: Trastuzumab SC (First SID, then Vial Formulation) (Experimental): Participants will start with 7 cycles of SC trastuzumab 600 mg administration via SID and after cross-over will receive 7 injections of trastuzumab 600 mg with assisted administration using a conventional syringe and needle (SC vial formulation).
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab IV or SC will be administered as described.
  Other Names: Herceptin
Drug: Paclitaxel — Paclitaxel will be administered in accordance with local hospital practice.
  Arms: Pre-Randomization (Trastuzumab IV)
Drug: Docetaxel — Docetaxel will be administered in accordance with local hospital practice.
  Arms: Pre-Randomization (Trastuzumab IV)

SUMMARY:
This multicenter study in participants with HER2-positive eBC will investigate participants' pain and discomfort of SC trastuzumab (Herceptin) administered either via a single-use injection device (SID) or via vial for manual administration using a hand-held syringe (SC vial). In total, participants will obtain at least 18 cycles/1 year of trastuzumab (4 cycles of intravenous [IV] and 14 cycles of SC trastuzumab).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Hormonal therapy allowed as per institutional guidelines
* Left ventricular ejection fraction (LVEF) of greater than or equal to (>/=) 55 percent (%) measured by echocardiography (ECHO) prior to first dose of trastuzumab
* HER2-positive disease immunohistochemistry (IHC) 3+ or in-situ hybridization (ISH) positive as determined in a local laboratory that is experienced/certified in HER2-expression testing using an accurate and validated assay
* Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast
* No evidence of residual, locally recurrent or metastatic disease after completion of surgery and chemotherapy, or during concurrent chemotherapy (neo-adjuvant or adjuvant)
* Participants who have completed all (neo)adjuvant treatment or participants after adjuvant chemotherapy with doxorubicin and cyclophosphamide (AC) to whom the 4 subsequent cycles of trastuzumab in combination with paclitaxel or docetaxel are indicated per local practice
* Not more than 3 months should have elapsed since the last dose of adjuvant chemotherapy in case of subsequent treatment scheme

Exclusion Criteria:

* Previous neoadjuvant or adjuvant breast cancer treatment with an approved or investigational anti-HER2 agent
* History of other malignancy that can affect compliance with the protocol or interpretation of results. Participants with curatively treated carcinoma in situ of the cervix or basal cell carcinoma, and participants with other curatively treated malignancies who have been disease-free for at least 5 years, are eligible. Participants with previous ductal carcinoma in situ (DCIS) of the breast are also eligible for the study
* Participants with severe dyspnea at rest or requiring supplementary oxygen therapy
* Participants with other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Prior maximum cumulative dose of doxorubicin >360 mg/m2 or maximum cumulative dose of epirubicin >720 mg/m2 or equivalent
* Serious cardiac illness or medical conditions that would preclude the use of trastuzumab, specifically: history of documented congestive heart failure (CHF), high-risk uncontrolled arrhythmias, angina pectoris requiring medication, clinically significant valvular disease, evidence of transmural infarction on electrocardiogram (ECG), diagnosed poorly controlled hypertension
* Known infection with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Pregnant or lactating women
* Concurrent enrollment in another clinical trial using an investigational anticancer treatment, including hormonal therapy, bisphosphonate therapy and immunotherapy, within 28 days prior to the first dose of study treatment
* Known hypersensitivity to trastuzumab, murine proteins, to any of the excipients of Herceptin®, or the adhesive of the SC device, or a history of severe allergic or immunological reactions, e.g., difficult to control asthma
* Inadequate bone marrow, hepatic, or renal function
* Major surgical procedure or significant traumatic injury within 14 days prior to the first dose of study treatment or anticipated need for major surgery during the course of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Participant Pain as Measured on a 10 Centimeter (cm) Visual Analogue Scale | Week 13 up to Week 52
Participant Discomfort as Measured on a 10 cm Visual Analogue Scale | Week 13 up to Week 52

SECONDARY OUTCOMES:
Healthcare Professional Satisfaction With SC Formulation as Assessed by Health Care Professional Questionnaire (HCPQ) | Week 22
Patient Satisfaction With SC Formulation as Assessed by Patients Satisfaction Questionnaire (PSQ) | Week 52
Healthcare Professional Perceived Time Savings With SC Trastuzumab as Assessed by HCPQ | Week 22
Percentage of Participants With Adverse Events | Baseline up to approximately 3 years
Overall Survival | From first study treatment to death from any cause, assessed up to approximately 4.5 years
Disease-Free Survival, Assessed as per Institutional Practice or American Society of Clinical Oncology (ASCO) Adjuvant Follow-up Guidelines 2006 | From first study treatment to documented disease progression or death, assessed up to approximately 3 years
Number of Days on Trastuzumab Treatment | Week 1 up to Week 52
Total Daily Dose of Trastuzumab | Week 1 up to Week 52
Cumulative Dose of Trastuzumab | Week 1 up to Week 52
Duration of Treatment | Week 1 up to Week 52
Duration of Safety Observation | 28 days after last study treatment (up to Week 56)
Duration of Follow-Up | 25 months after last study treatment (up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Belarus (4):
  - State Inst N.N. Alexandrov Republican Scientific & Practical Centre of Oncology & Medical Radiology, A/g Lesnoy, Minsk Region
  - Healthcare Institution "Brest Regional Oncologic Dispensary", Brest
  - Minsk City Clinical Oncologic Dispensary, Minsk
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Kazakhstan (3):
  - Kazakh Scientific Research Institution Of Oncology and Radiology; Chemotherapy department, Almaty
  - Almaty Cancer Hospital; Chemotherapy department, Almaty
  - Oncology centre of Astana; Chemotherapy department, Astana